CLINICAL TRIAL: NCT00303732
Title: PTK787/ZK222584 and RAD001 for Patients With Advanced Solid Tumors
Brief Title: Vatalanib and Everolimus in Treating Patients With Advanced Solid Tumors
Acronym: PTK/RAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel George, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012347; DUMC-6626-04-12R0 (Other: Duke IRB legacy number); CDR0000454988 (Other: National Cancer Institute)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus; vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTK787, RAD001 (Experimental): PTK787 (vatalinib) 1000 mg daily, RAD001 (everolimus) 5 mg daily
  Interventions: Drug: RAD001 (everolimus); Drug: PTK787 (vatalanib)

INTERVENTIONS:
Drug: RAD001 (everolimus)
  Other Names: Afinitor
Drug: PTK787 (vatalanib)

SUMMARY:
RATIONALE: Vatalanib and everolimus may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of vatalanib and everolimus and to see how well they work in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of vatalanib and everolimus in patients with advanced solid tumors.
* Determine the safety and tolerability of vatalanib and everolimus in patients with advanced solid tumors.
* Evaluate the safety and tolerability of vatalanib and everolimus at the MTD in patients with metastatic renal cell carcinoma (RCC).

Secondary

* Describe the non dose-limiting toxic effects associated with vatalanib and everolimus.
* Describe the pharmacokinetics of vatalanib and everolimus in patients with advanced solid tumors.
* Determine the functional extent of mTOR inhibition by changes in the phosphorylation status of S6K protein in peripheral blood mononuclear cells in patients treated with vatalanib and everolimus.
* Describe any clinical responses seen in patients with metastatic RCC in a dose-expansion cohort treated at the MTD.
* Observe overall survival of RCC patients treated with vatalanib and everolimus.
* Determine the time to progression of patients with RCC treated with vatalanib and everolimus.

OUTLINE: This is a phase I dose-escalation study followed by a phase Ib study.

* Phase I (solid tumors): Patients receive oral vatalanib on days 1-28 and oral everolimus on days 15-28 during course 1 and on days 1-28 during all subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of vatalanib and everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase Ib (renal cell carcinoma only): Patients receive oral vatalanib and oral everolimus at the MTD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor with radiographic evidence of metastatic disease

  * No standard therapy exists (phase I)
  * Unresectable or metastatic renal cell carcinoma (phase Ib)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* AST or ALT ≤ 2.5 times upper limit of normal (ULN)
* Total cholesterol < 300 mg/dL
* Triglycerides < 350 mg/dL
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance > 40 mL/min
* Negative proteinuria by dip stick OR total urinary protein ≤ 500 mg
* No uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with antihypertensive regimen
* No unstable angina pectoris
* No symptomatic congestive heart failure (New York Heart Association class III or IV heart disease)
* No uncontrolled serious cardiac arrhythmia (symptomatic supraventricular tachycardia or any ventricular tachycardia/fibrillation)
* No myocardial infarction in the past 6 months
* No uncontrolled diabetes
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No active or uncontrolled infection
* No uncontrolled hyperlipidemia
* No chronic renal disease
* No acute or chronic liver disease (e.g., hepatitis or cirrhosis)
* No impaired gastrointestinal (GI) function OR GI disease that may significantly alter the absorption of vatalanib or everolimus, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea and vomiting with solid food
  * Watery diarrhea > 5 times daily
  * Malabsorption syndrome
  * Bowel obstruction
  * Inability to swallow the tablets
* No confirmed HIV infection
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent severe and/or uncontrolled medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* No prior antivascular endothelial growth factor therapy
* More than 4 weeks since prior major surgery* (laparotomy)
* More than 2 weeks since prior minor surgery*
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* More than 6 weeks since prior antibody therapy
* More than 2 weeks since prior biologic/immunotherapy
* More than 2 weeks since prior limited-field radiotherapy
* More than 4 weeks since prior full-field radiotherapy
* More than 4 weeks since prior investigational agents
* Prior transfusions allowed provided blood counts are stable for > 2 weeks
* Concurrent epoetin alfa allowed
* No concurrent warfarin or similar oral anticoagulants that are metabolized by the cytochrome P450 system

  * Heparin and low molecular weight heparin allowed NOTE: *Insertion of a vascular access device is not considered major or minor surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-12; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of vatalanib and everolimus | Day 1 - 28
  Patients were evaluated on Day 1,14 and 28 for dose limiting toxicities
Safety and tolerability | Duration of study treatment
  Adverse events were assessed every 14 days for the length of the treatment period.
Safety and tolerability at the MTD in patients with metastatic renal cell carcinoma (RCC) | Duration of study treatment
  Patients were assessed for adverse events every 14 days while on study treatment

SECONDARY OUTCOMES:
Non dose-limiting toxicity | Duration of study treatment
  Patients were assessed every 14 days for non dose-limiting toxicity while on study treatment
Pharmacokinetics | Day 14 Cycle 1, Day 1 Cycle 2
  Blood was drawn for PK assessment on Day 14 of Cycle 1 and Day 1 of Cycle 2
Changes in the phosphorylation status of S6K protein in peripheral blood mononuclear cells | Day 1 and 28
  Samples were collected on Day 1 and at Day 28 of Cycle 1
Clinical response in patients with metastatic RCC | Duration of treatment
  patients underwent restaging studies every 2 cycles while on treatment for evidence of disease response
Overall survival of patients with RCC | Until death
Time to progression of patients with RCC | Duration of study treatment
  Patients were followed for evidence of disease progression as long as they remained on study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. George, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Speca JC, Mears AL, Creel PA, et al.: Phase I study of PTK787/ZK222584 (PTK/ZK) and RAD001 for patients with advanced solid tumors and dose expansion in renal cell carcinoma patients. [Abstract] J Clin Oncol 25 (Suppl 18): A-5039, 244s, 2007.